CLINICAL TRIAL: NCT01723592
Title: The Ability of an Orally Administered Preparation of Four Lactobacillus Species to Improve the Quality of the Vaginal Flora of Women With Breast Cancer and Chemotherapy. A Prospective Randomized Placebo-controlled, Double-blind Trial
Brief Title: Orall Administered Probiotics to Improve the Quality of the Vaginal Flora of Women With Breast Cancer and Chemotherapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Natural Resources and Life Sciences, Vienna, Austria (Other)
Responsible Party: Principal Investigator, Associate Prof. Ljubomir Petricevic MD, Assistant Professor, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: MUW EK 1417/2012
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2016-11

CONDITIONS: Breast Cancer
Keywords: chemotherapy; vaginal flora
MeSH Terms: conditions — Breast Neoplasms | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 30 participants in this group receive a oral lactose placebo
  Interventions: Dietary Supplement: Oral lactose placebo
- Probiotics (Active Comparator): 30 participants in this group receiving oral probiotic capsules for 7 days twice daily containing four lyophilised Lactobacillus strains belonging to the species:
  L.rhamnosus/ LbV96 (DSM 22560)
  L.jensenii /LbV 116 (DSM 22567)
  L.crispatus/ Lbv88 (DSM 22566)
  L.gasseri /LbV 150N (DSM 22583)
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics oral probiotic capsules for 7 days twice daily containing four lyophilised Lactobacillus strains,L.rhamnosus/ LbV96 (DSM 22560),L.jensenii /LbV 116 (DSM 22567),L.crispatus/ Lbv88 (DSM 22566),L.gasseri /LbV 150N (DSM 22583)
  Other Names: L.rhamnosus/ LbV96 (DSM 22560); L.jensenii /LbV 116 (DSM 22567); L.crispatus/ Lbv88 (DSM 22566); L.gasseri /LbV 150N (DSM 22583)
  Arms: Probiotics
Dietary Supplement: Oral lactose placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this study is the improvement of the vaginal flora by at least two grades of the Nugent scale after application of oral probiotics.

DETAILED DESCRIPTION:
The aim of this study is the improvement of the vaginal flora by at least two grades of the Nugent scale. Improvement of Nugent scores should be considered the primary end point of the study. The outcome of the study would be considered positive if significantly more women in the verum cohort achieve such improvement than in the placebo cohort.

ELIGIBILITY:
Inclusion Criteria:

Only women with breast cancer and neoadjuvant / adjuvant chemotherapy, at least 4 weeks postoperative, without vaginal bleeding without abnormal vaginal discharge, Only women with Nugent scores between 4 and 6

Exclusion Criteria:

Patients with diarrhoea, constipation, vaginal or urinary tract infection requiring antibacterial treatment and women receiving antibiotic therapy in the previous 4 weeks.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
change in Nugent score between baseline and end of treatment (improvement or no improvement) | day 0, 7 and day 14 of oral probiotic application
  Using Nugent scoring system, from each participant first swab from the vagina will be taken before start of oral probiotic use.(baseline information) Second swab will be taken on the day following the last administration.(information about change in Nugent)

SECONDARY OUTCOMES:
Isolation of specific Lactobacilli from vaginal microbiologic cultures after oral administration of probiotic | day 0, 7 and day 14 after oral probiotic application
  From each participant, a vaginal swab for microbiologic cultures will be taken on the first day and that following the last administration for Isolation of oral applied probiotic strains as well as non-lactobacilli-flora.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Kiss, MD, Study Director — Medical University of Vienna, Dept. of Obstetrics and Gynecology
Locations (1):
- Medical University of Vienna - Department of Obstetrics and Gynecology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No